CLINICAL TRIAL: NCT02059551
Title: Diagnostic Performances of Magnetic Resonance Imaging Combined With Venous Ultrasonography of the Legs for Pulmonary Embolism
Brief Title: Magnetic Resonance Imaging Combined With Venous Ultrasonography of the Legs for Pulmonary Embolism
Acronym: IRM-EP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120133
Record Dates: First submitted 2014-01-29; First posted 2014-02-11 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; magnetic resonance imaging; venous ultrasonography of the legs; diagnostic performances
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): In case of positive D-dimer testing or in patients with a high clinical probability of PE, these patients have MRI protocol combined with venous ultrasonography of the legs. MRI includes 2 different sequences: Unenhanced steady-state-free precession sequences (SSFP) sequences and angiography sequences. (please see \\\"intervention section\\\" for more details). MRI readings will be performed centrally by two independent readers blinded to the results of diagnostic reference standard. Venous ultrasonography of the legs will be interpreted locally.
  Interventions: Procedure: MRI combined with venous ultrasonography of the legs

INTERVENTIONS:
Procedure: MRI combined with venous ultrasonography of the legs — In case of positive D-dimer testing or in patients with a high probability of PE, MRI and a venous ultrasonography of the legs are done.MRI protocol includes 2 sequences: 1-Unenhanced steady-state-free precession sequences (SSFP) are acquired first without ECG-gating or breath-holding in the axial plane in the multiphase cine mode, with 6 phases per location.The acquisition is repeated to cover 2-3 of the thorax, from the roof of the aorta to the diaphragm. 2- A pulmonary gradient recalled echo (GRE) sequence is performed in the axial plane.The acquisition is triggered to start when contrast enhancement occurred in the right ventricle.Two acquisitions are necessary to cover the anatomy. For each acquisition, 0.15 mL kg-1 body weight of DOTAREM Gadolinium is injected at a rate of 3 mL s-1 followed by an injection of 15 mL of normal saline at 3 mL s-1.Venous ultrasonography of the legs: the examination consists of a real-time B-mode examination of the common femoral and popliteal veins.

SUMMARY:
Magnetic resonance imaging (MRI) represents a promising technique but can not be used as an alternative test to multidetector CT in patients with suspicion of pulmonary embolism (PE) due to its low sensitivity and high proportion of inconclusive MRI. The purpose of this study is to evaluate diagnostic performances of MRI combined with venous ultrasonography of the legs in patients with suspicion of PE.

ELIGIBILITY:
Inclusion criteria :

* age > or = 18 years
* clinical suspicion of PE
* Affiliate (e) to a social security
* provide written informed consent

Exclusion criteria :

* Unstable patient clinically in shock on arrival at the emergency department
* Current pregnancy
* Life expectancy less than 3 months (eg terminal cancer)
* Follow up at 3 months impossible
* Anticoagulation curative> 48 hours prior to inclusion
* Cons-indication to spiral chest CT: allergy to contrast or creatinine clearance below 30 ml / min calculated by the Cockcroft
* Cons-indication to MRI claustrophobia, presence of intraocular metallic implant or a pacemaker, an allergy to gadolinium, morbid obesity (weight> 130 kg, anteroposterior> 60 cm diameter)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
To assess diagnostic performances of MRI combined with venous ultrasonography of the legs in reference to Multi-Detector Computed Tomography and 3 months clinical follow-up | 51 months
  sensitivity, specificity, positive and negative likelihood ratios of the combination of MRI and venous ultrasonography of the legs

SECONDARY OUTCOMES:
To assess the diagnostic accuracy of a strategy combining clinical probability, D-dimer measurement, MRI and venous ultrasonography of the legs for PE | 51 months
  3-month thromboembolic events rate in patients who were left untreated on the basis of negative D-dimer measurement or negative combination of MRI + venous ultrasonography of the legs
To assess diagnostic performances of each MRI sequence combined or not to venous ultrasonography of the legs in reference to Multi-Detector Computed Tomography and 3 months clinical follow-up | 51 months
  sensitivity, specificity, positive and negative likelihood ratios of each MRI sequence (unenhanced 2D steady-state-free-precession (SSFP) and contrast-enhanced 3D angiographic MR sequences) combined or not to venous ultrasonography of the legs in reference to Multi-Detector Computed Tomography and 3 months clinical follow-up
inter-reader agreement for MRI | 51 months
  Kappa coefficient of concordance calculated on the diagnoses on MRI by two radiologists blinded to the diagnostic reference strategy (multidetector CT angiography and follow-up 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: SANCHEZ Olivier, MD, PhD, Principal Investigator — Université Paris Descartes; Sorbonne Paris Cité; Service de Pneumologie et Soins Intensifs, Hôpital Européen Georges POmpidou; AP-HP
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Revel MP, Sanchez O, Lefort C, Meyer G, Couchon S, Hernigou A, Niarra R, Chatellier G, Frija G. Diagnostic accuracy of unenhanced, contrast-enhanced perfusion and angiographic MRI sequences for pulmonary embolism diagnosis: results of independent sequence readings. Eur Radiol. 2013 Sep;23(9):2374-82. doi: 10.1007/s00330-013-2852-8. Epub 2013 May 8. PMID 23652845
- [Background] Revel MP, Sanchez O, Couchon S, Planquette B, Hernigou A, Niarra R, Meyer G, Chatellier G. Diagnostic accuracy of magnetic resonance imaging for an acute pulmonary embolism: results of the 'IRM-EP' study. J Thromb Haemost. 2012 May;10(5):743-50. doi: 10.1111/j.1538-7836.2012.04652.x. PMID 22321816
- [Background] Stein PD, Chenevert TL, Fowler SE, Goodman LR, Gottschalk A, Hales CA, Hull RD, Jablonski KA, Leeper KV Jr, Naidich DP, Sak DJ, Sostman HD, Tapson VF, Weg JG, Woodard PK; PIOPED III (Prospective Investigation of Pulmonary Embolism Diagnosis III) Investigators. Gadolinium-enhanced magnetic resonance angiography for pulmonary embolism: a multicenter prospective study (PIOPED III). Ann Intern Med. 2010 Apr 6;152(7):434-43, W142-3. doi: 10.7326/0003-4819-152-7-201004060-00008. PMID 20368649